CLINICAL TRIAL: NCT02532075
Title: The Effect of a Respiratory Muscle Warm-up Prior to Exercise in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: The Effect of a Respiratory Muscle Warm-up Prior to Exercise in Patients With Chronic Obstructive Pulmonary Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: University of Portsmouth (Other)
Responsible Party: Principal Investigator, Craig Williamson, PhD Research Student, University of Portsmouth
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: RWU-01
Record Dates: First submitted 2015-08-13; First posted 2015-08-25 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Respiratory Muscle Warm Up
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Inspiratory Warm Up (Experimental): (IWU). Two sets of 15 breaths
  Interventions: Other: Inspiratory Warm Up
- Expiratory Warm Up (Experimental): (EWU). Two sets of 15 breaths
  Interventions: Other: Expiratory Warm Up
- Combination Warm Up (Experimental): (RWU). One set of 15 breaths inspiratory and one set of 15 breaths expiratory
  Interventions: Other: Combination Warm Up
- Control Trial (Other): No warm up
  Interventions: Other: Control Trial

INTERVENTIONS:
Other: Inspiratory Warm Up — Inspiratory muscle warm up. Inhaling against a resistance for two sets of 15 breaths using a PowerLung.
  Arms: Inspiratory Warm Up
Other: Expiratory Warm Up — Expiratory muscle warm up. Exhaling against a resistance for two sets of 15 breaths using a PowerLung.
  Arms: Expiratory Warm Up
Other: Combination Warm Up — Combination of inspiratory and expiratory muscle warm up. One set of 15 breaths inhaling followed by one set 15 breaths exhaling.
  Arms: Combination Warm Up
Other: Control Trial — Control Trial. No respiratory muscle warm up to act as a comparison to the other three intervention trials.
  Arms: Control Trial

SUMMARY:
The purpose of this study is to investigate the effects of performing a breathing muscle warm up before exercise in patients who have chronic obstructive pulmonary disease (COPD). The main aim is to see whether performing a breathing muscle warm up can improve distance walked in a 6 minute walk test and also decrease perceptions of effort and breathlessness.

DETAILED DESCRIPTION:
The study will follow a counter-balanced repeated measures design involving six visits to the exercise laboratory. Following pre-screening and familiarisation (visits 1 and 2), participants will perform inspiratory warm up, expiratory warm up, combination warm up and control trials (visits 3 - 6) in a counter-balanced order separated by at least 48 hours between trials.

The four separate sessions will contain: lung function measurements assessed by performing breathing manoeuvres through a mouthpiece (spirometery or body plethysmography) before performing a breathing muscle warm up by breathing against a resistance through a small handheld device (PowerLung). Participants will then be asked perform a second set of lung function measurements and will then be asked to perform a 6 minute walk test wearing a face mask and a portable device (gas analysis), a small device clipped to a finger (pulse oximeter) and wearing a heart rate monitor. During this 6 minute walk test participants will also be asked to rate their perceived effort and level of breathlessness at 60m intervals. Following the test there will be a period of seated rest wearing the face mask and portable device for up to 20 minutes with one more set of lung function measurements.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of COPD
* Aged between 35 and 90 years
* Able to fluently read and speak English
* Willing and able to sign informed consent
* Be able to comply with the procedures outlined for the study

Exclusion Criteria:

* Cardiac disease (including arrhythmias)
* A medicinal requirement for rate limiting calcium antagonists or beta blockers
* Cerebrovascular disease
* Peripheral vascular disease
* Requirement for supplemental oxygen therapy
* CO2 (carbon dioxide) retention
* Malignancy
* Orthopaedic or neurological conditions effecting the ability to exercise
* Clinically apparent heart failure
* Renal, hepatic or inflammatory disease
* Instability of COPD
* Any other reason leading to the inability to complete the requirements of the study.

Additionally: If participants have a resting HR above 120beats.min-1, systolic blood pressure above 180mm Hg or diastolic blood pressure above 100mm Hg prior to the 6 minute walk test they will not be able to commence the test.

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-02; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Distance walked in the 6 minute walk test | Estimate is 4 weeks per participant to complete all trials. Measured during each trail that is expected to last 1-2 hours. (Trial format is described elsewhere).
Rating of perceived exertion (RPE) in the 6 minute walk test | Estimate is 4 weeks per participant to complete all trials. Measured during each trail that is expected to last 1-2 hours. (Trial format is described elsewhere).
  Measured from 1 minute pre 6 minute walk test to cessation of the test and at 60 metre intervals throughout.
Rating of dyspnoea during the six minute walk test | Estimate is 4 weeks per participant to complete all trials. Measured during each trail that is expected to last 1-2 hours. (Trial format is described elsewhere).
  Measured from 1 minute pre 6 minute walk test to cessation of the test and at 60 metre intervals throughout.

SECONDARY OUTCOMES:
Heart rate (HR) | Estimate is 4 weeks per participant to complete all trials. Measured during each trail that is expected to last 1-2 hours. (Trial format is described elsewhere).
  Measured from 1 minute pre 6 minute walk test to cessation of the test and at 60 metre intervals throughout.
Expired gas | Estimate is 4 weeks per participant to complete all trials. Measured during each trail that is expected to last 1-2 hours. (Trial format is described elsewhere).
  Measured from a few minutes prior to the six minute walk test until 20 minutes post test (or until VO2 returns to baseline following test). A brief gap in measurement will occur 5 minutes test to allow for a measure of pulmonary function.
Peripheral arterial oxygen saturation (SpO2) | Estimate is 4 weeks per participant to complete all trials. Measured during each trail that is expected to last 1-2 hours. (Trial format is described elsewhere).
  Measured from 1 minute pre 6 minute walk test to cessation of the test and at 60 metre intervals throughout.
Pulmonary function: maximal inspiratory mouth pressure (MIP) | Estimate is 4 weeks per participant to complete all trials. Measured during each trail that is expected to last 1-2 hours. (Trial format is described elsewhere).
  Measured pre respiratory warm up, post respiratory warm up and post 6 minute walk test (control trial will only be measured pre and post exercise test).
Pulmonary function: maximal expiratory mouth pressure (MEP) | Estimate is 4 weeks per participant to complete all trials. Measured during each trail that is expected to last 1-2 hours. (Trial format is described elsewhere).
  Measured pre respiratory warm up, post respiratory warm up and post 6 minute walk test (control trial will only be measured pre and post exercise test).
Pulmonary function: specific airway resistance (sRaw) | Estimate is 4 weeks per participant to complete all trials. Measured during each trail that is expected to last 1-2 hours. (Trial format is described elsewhere).
  Note: only if body plethysmography is available. Measured pre respiratory warm up, post respiratory warm up and post 6 minute walk test (control trial will only be measured pre and post exercise test).
Pulmonary function: airway resistance (Raw) | Estimate is 4 weeks per participant to complete all trials. Measured during each trail that is expected to last 1-2 hours. (Trial format is described elsewhere).
  Note: only if body plethysmography is available. Measured pre respiratory warm up, post respiratory warm up and post 6 minute walk test (control trial will only be measured pre and post exercise test).
Pulmonary function: functional residual capacity (FRCpleth) | Estimate is 4 weeks per participant to complete all trials. Measured during each trail that is expected to last 1-2 hours. (Trial format is described elsewhere).
  Note: only if body plethysmography is available. Measured pre respiratory warm up, post respiratory warm up and post 6 minute walk test (control trial will only be measured pre and post exercise test).
Pulmonary function: peak inspiratory flow (PIF) | Estimate is 4 weeks per participant to complete all trials. Measured during each trail that is expected to last 1-2 hours. (Trial format is described elsewhere).
  Measured pre respiratory warm up, post respiratory warm up and post 6 minute walk test (control trial will only be measured pre and post exercise test).
Pulmonary function: peak expiratory flow (PEF) | Estimate is 4 weeks per participant to complete all trials. Measured during each trail that is expected to last 1-2 hours. (Trial format is described elsewhere).
  Measured pre respiratory warm up, post respiratory warm up and post 6 minute walk test (control trial will only be measured pre and post exercise test).
Pulmonary function: forced expiratory flow at 25, 50 and 75% maximal vital capacity) (FEF 25, 50, 75) | Estimate is 4 weeks per participant to complete all trials. Measured during each trail that is expected to last 1-2 hours. (Trial format is described elsewhere).
  Measured pre respiratory warm up, post respiratory warm up and post 6 minute walk test (control trial will only be measured pre and post exercise test).
Pulmonary function: forced expiratory volume in one second (FEV1) | Estimate is 4 weeks per participant to complete all trials. Measured during each trail that is expected to last 1-2 hours. (Trial format is described elsewhere).
  Measured pre respiratory warm up, post respiratory warm up and post 6 minute walk test (control trial will only be measured pre and post exercise test).
Pulmonary function: forced vital capacity (FVC) | Estimate is 4 weeks per participant to complete all trials. Measured during each trail that is expected to last 1-2 hours. (Trial format is described elsewhere).
  Measured pre respiratory warm up, post respiratory warm up and post 6 minute walk test (control trial will only be measured pre and post exercise test).
Pulmonary function: residual volume (RV) | Estimate is 4 weeks per participant to complete all trials. Measured during each trail that is expected to last 1-2 hours. (Trial format is described elsewhere).
  Note: only if body plethysmography is available. Measured pre respiratory warm up, post respiratory warm up and post 6 minute walk test (control trial will only be measured pre and post exercise test).
Pulmonary function: tidal volume (VT) | Estimate is 4 weeks per participant to complete all trials. Measured during each trail that is expected to last 1-2 hours. (Trial format is described elsewhere).
  Measured pre respiratory warm up, post respiratory warm up and post 6 minute walk test (control trial will only be measured pre and post exercise test).
Pulmonary function: total lung capacity (TLC) | Estimate is 4 weeks per participant to complete all trials. Measured during each trail that is expected to last 1-2 hours. (Trial format is described elsewhere).
  Note: only if body plethysmography is available. Measured pre respiratory warm up, post respiratory warm up and post 6 minute walk test (control trial will only be measured pre and post exercise test).
Pulmonary function: inspiratory residual volume (IRV) | Estimate is 4 weeks per participant to complete all trials. Measured during each trail that is expected to last 1-2 hours. (Trial format is described elsewhere).
  Note: only if body plethysmography is available. Measured pre respiratory warm up, post respiratory warm up and post 6 minute walk test (control trial will only be measured pre and post exercise test).
Pulmonary function: expiratory residual volume (ERV) | Estimate is 4 weeks per participant to complete all trials. Measured during each trail that is expected to last 1-2 hours. (Trial format is described elsewhere).
  Note: only if body plethysmography is available. Measured pre respiratory warm up, post respiratory warm up and post 6 minute walk test (control trial will only be measured pre and post exercise test).
Pulmonary function: inspiratory capacity (IC) | Estimate is 4 weeks per participant to complete all trials. Measured during each trail that is expected to last 1-2 hours. (Trial format is described elsewhere).
  Measured pre respiratory warm up, post respiratory warm up and post 6 minute walk test (control trial will only be measured pre and post exercise test).
Pulmonary function: inspiratory vital capacity (IVC) | Estimate is 4 weeks per participant to complete all trials. Measured during each trail that is expected to last 1-2 hours. (Trial format is described elsewhere).
  Measured pre respiratory warm up, post respiratory warm up and post 6 minute walk test (control trial will only be measured pre and post exercise test).

CONTACTS AND LOCATIONS:
Overall Officials: Craig Williamson, MSc, Principal Investigator — PhD Research Student
Locations (1):
- University of Portsmouth - Department of Sport and Exercise Science, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No